CLINICAL TRIAL: NCT03396328
Title: Effects of Intensive Low-Salt Diet Education by Mobile Application on Albuminuria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2017-0906
Record Dates: First submitted 2018-01-04; First posted 2018-01-10 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Albuminuria
MeSH Terms: conditions — Albuminuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional education (Active Comparator)
  Interventions: Behavioral: conventional low salt education
- Low salt dietary education by smartphone application (Experimental)
  Interventions: Behavioral: Intensive low salt dietary education by smartphone application

INTERVENTIONS:
Behavioral: conventional low salt education — conventional low salt education
  Arms: Conventional education
Behavioral: Intensive low salt dietary education by smartphone application — Participants are provided with information on food and recipe, which allows them to record daily meals in their applications. Through the mobile application, the participants receive information on daily salt intake. Based on this information, the clinical nutritionist coach sets a goal for low salt diet and provides feedback to the patients through the mobile application. The clinical nutritionist coach checks the activity of the user more than twice a week and sends in-app messages to maintain compliance.
  Arms: Low salt dietary education by smartphone application

SUMMARY:
Albuminuria is a known risk factor for cardiovascular disease (CVD), chronic kidney disease (CKD) progression, all cause mortality. Inhibition of the renin-angiotension-aldosterone system (RAAS) plays an important role in the reduction of albuminuria and preservation of renal function in patients with CKD and it is known that the daily intakes of sodium have a significant effect on the activity of RAAS. Dietary sodium restriction has been shown to enhances the blood pressure, albuminuria, and renal function preservation. Furthermore, recent study has shown that intensive low-salt dietary education reduces albuminuria in patients with CKD. The average sodium intake of Koreans is 4,791 mg/d, which is higher than other countries. It is difficult for medical staff in Korea to invest enough time in low salt diet.

Recently, the development of health-related applications (apps) has been carried out worldwidely, and researches on lifestyle improvement using apps have been actively studied. However, there is no research yet on whether intensive education using an apps can affect lifestyle habits and thus changes in actual new features. Smartphone apps may provide an alternative to resource-intensive low salt diet-education. Therefore, this study aims to investigate the effect of intensive low salt diet training on the changes of albuminuria using application.

DETAILED DESCRIPTION:
This is an pen-label, case-control, randomized clinical trial.

* Run-in period (8 weeks) : before 8 weeks of study initiation, all of the patients have to stop all RAAS blockers or diuretics and switch to antihypertensive agents of other categories such as calcium channel blockers.
* 0-8 weeks : After run-in period, the patients complete laboratory examination and a dish frequency questionnaire. From 0 weeks, all participants will be prescribed valsartan 80mg per day until the end of study.
* 8-16 weeks : After 8 weeks, the patients will be randomly assigned to receive an low-salt dietary intervention after second laboratory examination.

Usual education : Conventional education at an outpatient clinic Intensive education : Low salt diet education through Smartphone app

The patients in the conventional education group will receive routine CKD education once at an outpatient clinic. Otherwise, the patients in the intensive education group will be trained low salt diet through smartphone app.

ELIGIBILITY:
Inclusion Criteria:

* Age : 19-65
* Underlying hypertension or antihypertensive medication , or Systolic blood pressure ≧ 140 mmHg or Diastolic blood pressure ≧ 90
* Modification of Diet in Renal Disease study (MDRD) eGFR ≧ 30 ml/min per 1.73m2
* Random urine albumin-to-creatinine ratio ≧ 30 mg/g
* Smartphone ownership

Exclusion Criteria:

* Age under 18 or over 66
* Uncontrolled hypertension (BP>160/110 mmHg)
* Pregnancy within 6 months
* Serum potasium > 5.5 mEq/L
* malignancy
* a diagnosis of CVD (cerebral infarction, hemorrhagic infarction, acute myocardial infarction or unstable angina, coronary angioplasty, or coronary artery bypass surgery) within the last 6 months
* Contraindication to angiotensin II receptor blocker
* life expectancy less than 6 months

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
Decrements of 24-hour urine albumin levels | 12 weeks after low salt diet education start
  Decrements of 24-hour urine albumin levels 12 weeks after low salt diet education

SECONDARY OUTCOMES:
Decrements of 24-hour urine sodium | 12 weeks after low salt diet education start
Change of blood pressure with a sphygmomanometer | 12 weeks after low salt diet education start

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Nephrology, Department of Internal Medicine Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No